CLINICAL TRIAL: NCT04837976
Title: Views and Priorities of Lifestyle Factors in the Management of Non-motor Symptoms in Parkinson's Disease: Qualitative Interviews and Consensus Workshops With Patients, Caregivers, and Healthcare Professionals
Brief Title: Lifestyle and Non-motor Symptom Management in Parkinson's Disease
Status: Terminated | Type: Observational
Why Stopped: Recruitment for the first stage has been completed. However the research team no longer has the staff or resources to complete stage 2 of the research.
Sponsor: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Sophie Lawrie, PhD Candidate, Oxford Brookes University
Other Study IDs: F.20.09.02
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Parkinson Disease; Fatigue
Keywords: Qualitative; Semi-structured interviews; Thematic analysis; Framework; Nominal Group Technique; Consensus methods
MeSH Terms: conditions — Parkinson Disease; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Individuals with Parkinson's Disease
  Interventions: Other: Semi-structured interviews and a consensus workshops using nominal group techniques.
- Supportive individuals: For example carers, family members or any other individual providing regular support or care to the person with Parkinson's.
  Interventions: Other: Semi-structured interviews and a consensus workshops using nominal group techniques.
- Healthcare Professionals
  Interventions: Other: Semi-structured interviews and a consensus workshops using nominal group techniques.

INTERVENTIONS:
Other: Semi-structured interviews and a consensus workshops using nominal group techniques. — Stage 1 of the study includes individual remote semi-structured interviews (one per participant). Stage 2 involves taking part in a consensus workshop with around 7 other Parkinson's experts, consisting of patients, supportive individuals and healthcare professionals.

SUMMARY:
Parkinson's Disease (PD) has generally been thought of as a movement disorder however other health-related symptoms, known as non-motor symptoms, are also very common. Non-motor symptoms can be very broad and present in numerous conditions, making identifying the symptoms of early-stage Parkinson's disease very difficult. Non-motor symptoms, including fatigue, and problems with sleep and mood, can happen decades before motor symptoms and have a greater impact on quality of life and psychological wellbeing. Despite this treatment options for non-motor symptoms are limited and therefore the development and testing of new treatments is a main priority.

Due to the limited treatments options available, self-management of symptoms through positive lifestyle changes is a warranted area of research. The perspectives amongst patients, caregivers, and HCP's regarding lifestyle behavior change and its impact on fatigue and related non-motor symptoms has yet to be investigated in detail. This study includes two stages: telephone interviews and online consensus workshops. Patients with PD whom have experience of fatigue, partners/caregivers and Healthcare professionals will be able to participate in interviews only, workshops only or both. The interviews will investigate patients, partners/caregivers and Healthcare Professionals views and priorities of lifestyle factors in the management of non-motor symptoms in Parkinson's disease as well as identifying factors that influence lifestyle changes amongst PD patients. Stage 2 will involve small consensus workshops to generate ideas and feedback related to the design and content of the soon-to be developed lifestyle program. Results from both stages of this study will be used to help develop and design a lifestyle management program for fatigue and associated non-motor symptoms in Parkinson's Disease.

DETAILED DESCRIPTION:
Global aim: To assess stakeholders (patients, supportive individuals, and HCP's) views and priorities of lifestyle factors in the management of fatigue and related non-motor symptoms in Parkinson's disease, in addition to identifying facilitators and barriers to lifestyle-related behavior change, in order to inform the development of a subsequent lifestyle intervention.

The study consists of two stages:

1. Semi-structured interviews (lasting around 60 minutes)
2. Online consensus workshops using a nominal group technique (2x 60 minute sessions)

Setting: Both stages will be conducted remotely. For Stage 1 interviews will be conducted over the telephone (with or without videoconferencing). Stage 2 will use an online brainstorming platform to run the consensus workshop with concurrent videoconferencing.

Participants: For both stages' participants will include individuals with Parkinson's Disease, supportive individual's (partners/caregivers/family members/significant others) and healthcare professionals.

Analysis:

Stage 1- Interviews will be analyzed using thematic analysis and framework mapping onto the COM-B model. Themes will be deductively mapped onto the categories and its associated constructs of the Capability, Opportunity and Motivation to Behaviour (COM-B) model to identify specific targetable aspects of behavior that may need to be addressed in the subsequent lifestyle intervention. A secondary categorical form narrative analysis of the interviews will also be conducted to supplement the main group analysis by providing a detailed insight into the experiences and stories of participants in relation to lifestyle changes on an individual level.

Stage 2- Responses during the consensus workshop will be analyzed using frequency counts and descriptive. Data will include a complete list of ideas, scores allocated to each idea, the overall rank of each idea and any additional comments made by participants.

ELIGIBILITY:
Inclusion criteria

A) Patients

* A diagnosis of idiopathic Parkinson's Disease
* Age of 18 years or above
* Current or previous experience of persistent fatigue
* Able to communicate clearly in English over the telephone/online for over an hour
* Have access to a working computer and internet connection (required for stage 2 only).

B) Supportive person (partner/family member/caregiver)

* Age of 18 years or above
* A supportive person of an individual with Parkinson's Disease whom has already consented to take part in the research. Supportive individuals cannot take part without an associated individual with Parkinson's Disease having already consented.
* Has regular contact with and is involved in the care and/or support of an individual diagnosed with Idiopathic Parkinson's Disease.
* Able to communicate clearly in English over the telephone/online for over an hour
* Have access to a working computer and internet connection (required for stage 2 only).

C) Healthcare Professionals

* Healthcare Professional with at least 2 years experience of Parkinson's disease treatment/management/clinical care and/or an academic currently working in the area of Parkinson's Disease treatment.
* Have access to a working computer and internet connection (required for stage 2 only).

Exclusion criteria

A) Patients

* Reduced cognition that would preclude active involvement and capacity to consent to participate
* Unable to communicate clearly in English over the telephone/online for over an hour.

B) Partners/Caregivers

* Reduced cognition that would preclude active involvement and capacity to consent to participate
* Unable to communicate clearly in English over the telephone/online for over an hour.

C) Health Care Professional

* Less than 2 years' experience in the treatment/management/clinical care of individuals with Parkinson's disease as determined by self-report
* They have worked in this field but have stopped for two years or more.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and Supportive Individuals will be recruited from a Neurology clinic at Oxford University Hospitals NHS Foundation Trust (OUHFT) and from the Parkinson's UK website. Healthcare proffesionals will be recruited via the Parkinson's UK Excellence Network.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Themes related to the views and priorities of lifestyle factors in relation to fatigue and non-motor symptom management in Parkinson's Disease. | Assessed during the interview (60 minutes) after enrollment
Facilitators to dietary and exercise-based lifestyle change amongst patients with Parkinson's disease. | Assessed during the interview (60 minutes) after enrollment
Barriers to dietary and exercise-based lifestyle change amongst patients with Parkinson's disease. | Assessed during the interview (60 minutes) after enrollment
Identified behavioral targets for the intervention as indicated by the mapping of themes onto the COM-B model (capability, opportunity or motivation) | Assessed during the interview (60 minutes) after enrollment
A list of potential methods of intervention delivery, structure and content, ranked in order of preference created during consensus workshops. | From participation in the first consensus session after enrollment until session 2 (around 1-2 weeks later)

OTHER OUTCOMES:
Parkinson's Fatigue Scale (PFS-16) | Once prior to the interview and/or consensus workshop.
  A patient-rated scale that measures fatigue in Parkinson's disease ranging from 0 to 80.. A Score of 8 or above indicates the presence of significant fatigue. Higher scores correspond to worse fatigue.
Becks Depression Inventory (BDI-II) | Once after enrollment, prior to the interview- patients only
  A 21-item self-reported questionnaire with scores for each item ranging from 0 (absence of symptoms) to 3 (severe symptoms). Total scores range between 0 and 63 with higher scores indicating greater severity of depressive symptoms.
Geriatric Anxiety Scale (GAS) | Once after enrollment, prior to the interview- patients only
  Self-reported assessment of anxiety symptoms amongst older adults. Scores range from 0 to 20, with scores of 0-8 indicating an absence of clinically significant anxiety and scores of 9 and above indicating the presence of clinically significant anxiety.
Apathy Evaluation Scale (AES) | Once after enrollment, prior to the interview- patients only
  Self-reported assessment of apathy symptoms. The total AES score ranges between 18 to 72 with a lower score indicating greater apathy.
Parkinson's Disease Sleep Scale (PDSS-2) | Once after enrollment, prior to the interview- patients only.
  Self-rated assessment to quantify the level of sleep disruption in Parkinson's Disease. Scores range from 0 to 60, with higher scores representing more severe nocturnal disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Lawrie, Principal Investigator — Oxford Brookes University
Locations (1):
- Oxford Brookes University, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No